CLINICAL TRIAL: NCT04025892
Title: A Pilot and Feasibility Study of Daily Weight Tracking to Manage Gestational Weight Gain During Pregnancy
Brief Title: Pregnancy Tracking Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate resources to support study start-up
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102563
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-05

CONDITIONS: Gestational Weight Gain
Keywords: pregnancy; digital health; daily weighing
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracking group (Experimental): Participants will be asked to track weight daily for six weeks
  Interventions: Behavioral: Daily weighing

INTERVENTIONS:
Behavioral: Daily weighing — Participants will be asked to use the scale to track their body weight daily at home for six weeks. They will receive a weekly email contact with weight change feedback and either a nutrition or physical activity tip for the week. The study procedures represent minimal risks, and participants will be reminded and encouraged to maintain their regular prenatal care contacts with their provider.

SUMMARY:
This pilot study will examine perceptions about daily weighing for pregnant women with overweight or obesity by testing the feasibility, acceptability, and preliminary efficacy of daily weighing for reducing excess gestational weight gain (GWG) within the context of a low intensity, digital-health based intervention delivered remotely with electronic feedback to participants.

ELIGIBILITY:
Inclusion Criteria:

* women ages 18-34
* first pregnancy and at 13-20 weeks' gestation
* low-risk uncomplicated pregnancy
* overweight or obese at the time they became pregnant
* willing to receive emails.

Exclusion Criteria:

* Individuals who are not pregnant
* not willing to receive emails
* pregnant women expecting more than a single birth,
* outside the window of 13-20 weeks' gestation
* high-risk or complicated pregnancy for which participation would be contraindicated
* advanced maternal age according to obstetric guidelines (i.e., age 35 or older)
* diabetes
* history of eating disorders
* pre-pregnancy weight less than 25 kg/m2or greater than 36 kg/m2 (either not overweight or with extreme obesity)

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of scale use | Approximately 6 weeks
  The number of times weight is measured on the scale

SECONDARY OUTCOMES:
Weight change trajectories during scale use | Approximately 6 weeks
  Average weight change over the study duration
Knowledge of gestational weight gain guidelines | During baseline visit (~ 1 hour)
  Score of response from baseline survey item inquiring about awareness of gestational weight gain where greater score indicates greater knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Dori Steinberg, Principal Investigator — DUSON
Locations (1):
- Duke Global Digital Health Science Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No